CLINICAL TRIAL: NCT05731349
Title: Early Sepsis Care With the National Early Warning Score 2-guided Sepsis Hour-1 Bundle in the Emergency Department: A Hybrid Type 1 Effectiveness-Implementation Pilot Stepped Wedge Randomised Controlled Trial (NEWS-1 Trial Pilot Study)
Brief Title: Impact of Early Sepsis Care Guided by the National Early Warning Score 2 in the Emergency Department
Acronym: NEWS-1-TRIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Pamela Youde Nethersole Eastern Hospital (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other); Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Lam Pui Kin, Associate Professor of Emergency Medicine Practice, Department of Emergency Medicine, School of Clinical Medicine, Li Ka Shing Faculty of Medicine, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Project No. 19201161
Record Dates: First submitted 2023-01-26; First posted 2023-02-16 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; National Early Warning Score; Surviving Sepsis Campaign Hour-1 Bundle; Emergency Department; Implementation Sciences
MeSH Terms: conditions — Sepsis; Shock, Septic; Emergencies

STUDY DESIGN:
Intervention Model Description: Stepped-wedge, cluster-randomized trial
Masking Description: Masking is not feasible given the study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEWS-1 care (Experimental): During the interventional period, the 2018 Sepsis Hour-1 Bundle will be initiated in the ED if NEWS2 score ≥ 5.
  Interventions: Other: 2018 Surviving Sepsis Campaign Hour-1 Bundle
- Standard care (No Intervention): During the standard care period, emergency physicians will assess the patients based on history, physical examination, laboratory tests, chest radiography or other imaging studies, and will offer treatment based on clinical expertise, intuition, and local or international guidelines

INTERVENTIONS:
Other: 2018 Surviving Sepsis Campaign Hour-1 Bundle — 1. Measure lactate
  2. Obtain blood cultures before administering antibiotics
  3. Administer broad-spectrum antibiotics based on local guidelines
  4. Begin fluid resuscitation with up to 30 mL/kg crystalloid for hypotension or lactate level ≥ 4 mmol/L.
  5. Apply vasopressors if hypotensive during or after fluid resuscitation to maintain the MAP ≥ 65 mm Hg
  Arms: NEWS-1 care

SUMMARY:
The goal of this pilot clinical trial is to determine the feasibility of conducting a fully powered type 1 hybrid effectiveness-implementation trial on early sepsis care that is guided by early warning score in adult emergency department (ED) patients who have infection. The main questions it aims to answer are:

* Is it feasible to execute the trial procedure and fulfill the progression criteria to a full-scale trial?
* Does the Surviving Sepsis Campaign (SSC) Hour-1 Bundle care reduce the mortality of adult ED patients with a clinical diagnosis of infection and a National Early Warning Score 2 (NEWS2) equal to or greater than 5?
* What are the barriers to and facilitators of the implementation of the SSC Hour-1 Bundle in the ED settings?

Participants will receive the following SSC Hour-1 Bundle care during the intervention period:

* Blood lactate level measurement
* Blood cultures collection before administering antibiotics
* Broad-spectrum antibiotics
* Intravenous fluid
* Vasopressors if the blood pressure remains low during or after fluid replacement to maintain the mean arterial blood pressure equal to or greater than 65 mmHg

Researchers will compare patients who receive SSC Hour-1 Bundle triggered by a NEWS2 equal to or greater than 5 and patients who receive standard treatment based on clinical judgement to see if the SSC Hour-1 that is triggered by a high NEWS2 score could reduce mortality of adult ED patients with infection.

DETAILED DESCRIPTION:
Despite international endorsement and promulgation, the uptake of the sepsis-care bundles remains low across health-care settings. In most cases, clinicians are still offering sepsis care based on individual clinical judgement, intuition, skills, and available time and resources, leading to a variable standard of care at best and a suboptimal patient outcome in many cases. Significant knowledge gaps exist in the real-world effectiveness of sepsis bundles that are objectively triggered by the early warning score and in the best implementation strategy of sepsis bundle in the ED setting.

The sepsis care model in which the SSC Hour-1 Bundle is triggered objectively by a high NEWS2 score (≥ 5) (known as "NEWS-1 care" in this study) will be evaluated in this study. This pilot study is a type 1 hybrid effectiveness-implementation study, which contains all the major components of a planned full-scale hybrid trial intended to involve a larger sample size from more local EDs. This pilot study has two essential components:

First, the effectiveness component will evaluate the effect of the SSC Hour-1 Bundle in reducing 30-day all-cause mortality in adult patients presenting to the ED with a clinical diagnosis of infection and a NEWS2 ≥ 5. A prospective, stepped-wedge, cluster-randomized trial, which combines elements of a standard cluster-randomized design (intervention applied in clusters) and a before-after design (in which each cluster switches to the intervention), will be conducted in four EDs in Hong Kong. All study sites will start with an initial period of standard care; they will then switch in random order at intervals of two months to the NEWS-1 care in a unidirectional fashion until all hospitals have crossed over. Recruitment will continue in all study sites until the end of the trial.

Second, the implementation component will use a mixed-methods design to evaluate the uptake of the SSC Hour-1 Bundle using the Reach Effectiveness Adoption Implementation Maintenance (RE-AIM) framework, and determine the barriers to and facilitators of its implementation in daily practice.

The primary outcome of this pilot study is the feasibility of a full-scale type 1 hybrid trial on the NEWS-1 care, which will be determined based on the 14 pre-defined progression criteria to assess the feasibility of emergency staff in multiple centres to screen, recognise and recruit patients with suspected sepsis and to execute trial procedures; the feasibility of trial methods to decide whether a fully-powered trial should be undertaken to determine the safety and effectiveness of the intervention; and the feasibility of research staff to conduct the implementation evaluation. Please refer to the published study protocol for the 14 progression criteria.

We will not proceed to a full-scale trial if there is clear evidence of significant harm (safety criterion) or effect (equipoise criterion). As for the other progression criteria, no weighing will be added during evaluation and they will be considered collectively as we conclude the study.

ELIGIBILITY:
Inclusion Criteria:

ED patients aged ≥ 18 years who fulfil ALL of the following criteria:

* a clinical diagnosis of infection made by the treating emergency physicians
* require hospital admission
* a NEWS2 ≥ 5

Exclusion Criteria:

* age < 18 years
* currently pregnant
* neutropenic or post-chemotherapy fever, for which ED protocols for early antibiotics apply
* an advanced directive with a ceiling-of-care
* refusal of consent/pre-existing mental illness rendering consent impossible
* refusal of hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
All-cause 30-day mortality (in full-scale stepped wedge RCT) | 30 days
  The number of patients who die over 30 days

OTHER OUTCOMES:
All-cause in-hospital mortality (in full-scale stepped wedge RCT) | From the date of recruitment until the date of death from any cause or date of hospital discharge, whichever comes first, assessed up to 90 days
  The number of patients who die during the index hospitalization
All-cause 90-day mortality (in full-scale stepped wedge RCT) | 90 days
  The number of patients who die over 90 days
Sepsis-related in-hospital mortality (in full-scale stepped wedge RCT) | From the date of recruitment until the date of death from sepsis or date of hospital discharge, whichever comes first, assessed up to 90 days
  The number of patients who die during the index hospitalization because of sepsis, as judged by an independent emergency physician and an infectious disease specialist based on review of clinical notes and autopsy findings, if available
Intensive care unit admission (in full-scale stepped wedge RCT) | From the date of recruitment until the date of first documented intensive care unit admission or date of hospital discharge or date of death, whichever comes first, assessed up to 90 days
  Number of participants who require intensive care unit admission during the index hospitalization
Ventilator-free days over 30 days (in full-scale stepped wedge RCT) | Over 30 days following recruitment
  The number of ventilator-free days over 30 days after recruitment
The need for renal replacement therapy (in full-scale stepped wedge RCT) | From the date of recruitment until the date of first documented renal replacement therapy or date of hospital discharge or date of death, whichever comes first, assessed up to 90 days
  The number of patients who require renal replacement therapy during the index hospitalization that is not due to pre-existing renal failure
The total length of stay in the emergency department (in full-scale stepped wedge RCT) | From the time of emergency department registration to the time of check out from the emergency department or time of death in the emergency department, whichever comes first, assessed up to 7 days
  The total number of hour of patient stay in the emergency department
The total length of stay in the intensive care unit (in full-scale stepped wedge RCT) | From the date of intensive care unit admission until the date of discharge from the intensive care unit or date of death, whichever comes first, assessed up to 90 days
  The total number of days of patient stay in the intensive care unit
The total length of stay in the general ward (in full-scale stepped wedge RCT) | From the date of hospital admission to general ward until the date of hospital discharge or date of transfer out of general ward or date of death, whichever comes first, assessed up to 90 days
  The total number of days of patient stay in the general ward
The time to surgery (in full-scale stepped wedge RCT) | From the of emergency department registration until the first documented time of surgery or time of hospital discharge or time of death, whichever comes first, assessed up to 90 days
  The number of hours from ED registration to the first surgery for cases who receive surgery during the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Pui Kin Lam, MBBS, MPH, Principal Investigator — The University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Accident and Emergency Department, Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Accident and Emergency Department, Prince of Wales Hospital, Hong Kong
  - Accident and Emergency Department, Queen Mary Hospital, Hong Kong
  - Accident and Emergency Department, Tuen Mun Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be available on reasonable request 9 months after publication of the main results, subject to the additional research ethics approval on data sharing. Requests for data should be sent to lampkrex@hku.hk.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 9 months after publication of the main results
Access Criteria: De-identified study data will be available on reasonable request 9 months after publication of the main results, subject to the additional research ethics approval on data sharing.

REFERENCES:
- [Background] Lam RPK, Hung KKC, Lui CT, Kwok WS, Lam WWT, Lau EHY, Sridhar S, Ng PYT, Cheng CH, Tsang TC, Tsui MSH, Graham CA, Rainer TH. Early sepsis care with the National Early Warning Score 2-guided Sepsis Hour-1 Bundle in the emergency department: hybrid type 1 effectiveness-implementation pilot stepped wedge randomised controlled trial (NEWS-1 TRIPS) protocol. BMJ Open. 2024 Feb 1;14(2):e080676. doi: 10.1136/bmjopen-2023-080676. PMID 38307529